CLINICAL TRIAL: NCT04964102
Title: Associations of Communication Skills Workshop and Improvements in Stress, Burnout and Empathy and Psychometric Properties of Chinese Version of Perceived Stress Scale, Professional Fulfillment and Burnout Scale and Empathy Among Health Care Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-I Wu, Principal Investigator, Mackay Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20MMHIS092e
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Stress
Keywords: Professional burn out; Communication skills; empathy; fulfillment
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Workshop (Experimental): Workshop of Enhancing Interpersonal Effectiveness, Emotional Regulation and Clinical Communication Skills
  Interventions: Behavioral: Workshop of Enhancing Interpersonal Effectiveness, Emotional Regulation and Clinical Communication Skills

INTERVENTIONS:
Behavioral: Workshop of Enhancing Interpersonal Effectiveness, Emotional Regulation and Clinical Communication Skills — Workshop of Enhancing Interpersonal Effectiveness, Emotional Regulation and Clinical Communication Skills

SUMMARY:
This study aims to explore associations of burn out, stress, communication skills, interpersonal effectiveness and empathy level using data collected in pre and post assessments from "Workshop of Enhancing Interpersonal Effectiveness, Emotional Regulation and Clinical Communication Skills".

DETAILED DESCRIPTION:
The medical community is paying more and more attention to the nature of burnout, physiological, or physical stress of health care professionals (HCP). Burn out and stress not only affects the HCP themselves, but subsequently their team members, medical institutions, and patients. Recent research has found that HCP's stress, burnout, and dissatisfaction with work are associated with their practice time and leaving the job; as well as declines in quality of care, poor patient results, and medical errors.

There seems to be a two-way correlation between burn out and empathy. On the one hand, the more burn out, the lower the degree of empathy; on the other hand, the deficits in perspective substitution seems to be a risk factor for burn out. The increase in multiple perspectives and empathic attention seems prevent burn out. Other studies found that practicing clinical communication skills through practices and role-plays, and using emotional regulation methods to enable participants to express their attitudes and feelings about communicating difficult problems may help HCP improve their degree of empathy and communication skills. When such communication courses add combinations of stress management and social skills training can not only improve communication skills, increase empathy, but also prevent burnout and exhaustion.

Therefore, this study aims to explore associations of burn out, stress, communication skills, interpersonal effectiveness, and empathy level using data collected in pre- and post- assessments from 'Workshops of Enhancing Interpersonal Effectiveness, Emotional Regulation, and Clinical Communication Skills'. Before and after the workshop, information regarding HCP's burn out, perceived stress, empathy level, and interpersonal effectiveness will be assessed in order to understand whether the workshop has reached its goals and teaching effectiveness. All information regarding personal data will be de-identified and encrypted. These assessments are designed to evaluate the effectiveness of teaching activities in a general teaching environment. This study will also focus on the reliability and validity analysis of the short form research measures which used. It will conduct validation studies comparing the Chinese version of the measures which used with internationally well known but long research measures to make sure the reliability and validity. If these shorter forms have well validity, it may be able to use the short and simplified questionnaires for related research in the future.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 65 years old
* willing to attend the workshop and willing to participate this study

Exclusion Criteria:

* age less than 20 or over 65 years old

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS) Score before and after workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  The PSS scores is a rating tool used to gauge the course of stree. The minimum total score possible is 0 and the maximum total score possible is 40. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Differences in Empathy Scale before and after workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  The Empathy Scale is one of the first measures to achieve widespread use, contains four separate dimensions: social self-confidence, even-temperedness, sensitivity, and nonconformity. The instrument is scored on a scale of 0 (being the least empathetic possible) to 80 (being the most empathetic possible).
Differences in Insomnia Severity index (ISI) before and after workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  The ISI is a rating tool used to gauge of sleeping. Higher values represent a worse outcome.
Differences in the State and Trait Anxiety Index (STAI) before and after the workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Differences in Generalized Anxiety Disorder 7-item (GAD-7) before and after the workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  Self-administered 7 item instrument that uses some of the DSM-V criteria for GAD (General Anxiety Disorder) to identify probable cases of GAD along with measuring anxiety symptom severity. It can also be used as a screening measure of panic, social anxiety, and PTSD. It was modeled after the PHQ9 to be used quickly and effectively within a primary care setting.
Differences in Patient Health Questionnaire-9 (PHQ-9) before and after the workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Differences in Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) before and after the workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF; Endicott et al,1993). The Q-LES-Q-SF evaluates general activities that are assessed in the longer form of the Q- LES-Q. Each item uses a 5-point scale ranging from 1 (very poor) to 5 (very good). A total score is derived from 14 items with a maximum score of 70 and with higher scores indicating greater life satisfaction and enjoyment.
Differences in Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL) before and after the workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  Differences in Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL) may have coped with stressful events in life. The Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL) is a 59-item self-report scale designed to assess participants' use of DBT skills (e.g., acceptance, cognitive reappraisal, problem-solving) and maladaptive coping responses. The DBT-WCCL is a checklist designed to gauge ways of coping. As subjects go through the 59 questions, they can think about and evaluate different ways in which they may have coped with stressful events in life. Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL) effective coping subscale. Minimum score: 0. Maximum score: 3. Higher score indicates more frequent use of adaptive coping strategies. Lower score indicates less frequent use of adaptive coping strategies.
Differences in Jefferson Scale of Empathy (JSE) before and after the workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  The Jefferson Scale of Empathy (JSE) is to measure empathy in physicians, and other health professionals involved in patient care in a clinical setting; as well as students studying medicine and other forms of health care in preparation for working in a clinical setting. The minimum and maximum scores for JSE-HPS can be reached to 20 and 140, respectively. The more the higher scores indicate more empathic aspect or vice versa.
Differences in Interpersonal Reactivity Index (IRI) before and after the workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  The Interpersonal Reactivity Index (IRI) is a published measurement tool for the multi-dimensional assessment of empathy. 28 items using 5-point scales (A = does not describe me well to E = describes me very well) Sub-scales 4 sub-scales, each with 7 items: Fantasy assesses the extent to which individuals identify with fictional characters.
  Perspective-taking assesses the extent to which individuals spontaneously (try to) adopt others' points of view.
  Empathetic concern assesses the extent of individuals' "feelings of warmth, compassion, and concern for others." Personal distress assesses the extent of individuals "feelings of anxiety and discomfort" as a result of "another's negative experience." scores would range from 28 to 140
Differences in Maslach Burnout Inventory (MBI) before and after the workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  The Maslach Burnout Inventory (MBI) is a psychological assessment instrument comprising 22 symptom items pertaining to occupational burnout. All MBI items are scored using a 7 level frequency ratings from "never" to "daily." The MBI has three component scales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout. Scales should not be combined to form a single burnout scale. Maslach, Jackson, and Leiter[1] described item scoring from 0 to 6. There are score ranges that define low, moderate and high levels of each scale based on the 0-6 scoring.
Differences in Professional Fulfillment Index (PFI) before and after the workshop and Week 24 Assessed | Before and after workshop and 24 weeks
  Professional Fulfillment Index (PFI) is a 16-item instrument to assess physicians' professional fulfillment and burnout, designed for sensitivity to change attributable to interventions or other factors affecting physician well-being. All burnout items are scored on a 5-point Likert scale with options ranging from "not at all" to "extremely" for burnout items and "not at all true" to "completely true" for professional fulfillment items. Aggregate scores for burnout and professional fulfillment were calculated using the published approach, with possible scores ranging from 0 to 40 and 0 to 24, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan